CLINICAL TRIAL: NCT04565015
Title: An Open-Label, Single-Arm, Historically Controlled, Prospective, Multi-Center Phase III Study to Evaluate the Pharmacokinetics and Safety of Immune Globulin Intravenous (Human) GC5107 in Pediatric Subjects With Primary Humoral Immunodeficiency
Brief Title: Study of Immune Globulin Intravenous (Human) GC5107 in Pediatric Subjects With Primary Humoral Immunodeficiency
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: GC Biopharma Corp (Industry)
Collaborators: Atlantic Research Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GC5107D
Record Dates: First submitted 2020-09-07; First posted 2020-09-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Primary Immune Deficiency
MeSH Terms: conditions — Primary Immunodeficiency Diseases | interventions — gamma-Globulins; Fluid Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- GC5107 (Experimental): Immune Globulin Intravenous (Human), 10% Liquid
  Interventions: Biological: GC5107

INTERVENTIONS:
Biological: GC5107 — Intravenously infused at a dose of 300 - 900 mg per kg (of body weight) every 21 or 28 days for 12 months
  Other Names: GCC 10% IGIV; Immune Globulin Intravenous (Human), 10% Liquid

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics and safety of Immune Globulin Intravenous (Human) GC5107 in pediatric subjects with Primary Humoral Immunodeficiency (PHID).

DETAILED DESCRIPTION:
This is a prospective, open-label, single-arm, historically controlled, multi-center Phase III study to assess the pharmacokinetics and safety of Immune Globulin Intravenous (Human) GC5107 in pediatric subjects aged ≥ 2 years and < 17 years with PHID.

Subjects will receive intravenous infusions of the investigational product at the same dose and interval as used for their previous Immunoglobulin intravenous (IGIV) maintenance therapy. GC5107 will be infused every 21 or 28 days for a period of 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be ≥ 2 to < 17 years of age, at the time of signing the informed consent
* Pediatric subject has a confirmed and documented clinical diagnosis of Primary Humoral Immunodeficiency, including hypogammaglobulinemia or agammaglobulinemia
* Subject who has received 300 - 900 mg/kg of IGIV therapy at 21 or 28 day intervals for at least 3 months prior to this study
* Subject who has at least 2 documented plasma IgG trough level of ≥ 500 mg/dL at two infusion cycles (21 or 28 days) within 12 months prior to enrollment
* Subject who is willing to comply with all requirements of the protocol

Exclusion Criteria:

* Subject who has a history of clinically significant reactions or hypersensitivity to IGIV or other injectable forms of IgG
* Subject who has IgA deficiency and is known to have antibodies to IgA
* Subject who has secondary immunodeficiency
* Subject who has participated in another clinical study (other than an IGIV study) within 3 weeks prior to screening
* Subject who has been diagnosed with dysgammaglobulinemia or isolated IgG subclass deficiency or isolated IgA deficiency, or who has clinically significant impairment of cellular or innate immunity at the discretion of the Investigator
* Subject who has received blood products other than human albumin or human immune globulin within 6 months prior to enrollment

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2020-12-21 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
The Pharmacokinetic (PK) Plasma concentration-time curve of total IgG | before and after 5th infusion (12 or 16 weeks)
The Pharmacokinetic (PK) Half-life of total IgG | before and after 5th infusion (12 or 16 weeks)
The Pharmacokinetic (PK) Area under the curve of total IgG | before and after 5th infusion (12 or 16 weeks)
The Pharmacokinetic (PK) Volume of distribution of total IgG | before and after 5th infusion (12 or 16 weeks)
The Pharmacokinetic (PK) Maximum concentration of total IgG | before and after 5th infusion (12 or 16 weeks)
The Pharmacokinetic (PK) Minimum concentration of total IgG | before and after 5th infusion (12 or 16 weeks)
The Pharmacokinetic (PK) Time of maximum concentration of total IgG | before and after 5th infusion (12 or 16 weeks)
The Pharmacokinetic (PK) Clearance of total IgG | before and after 5th infusion (12 or 16 weeks)
Trough serum total IgG levels before each infusion of GC5107 in all subjects and the interval between infusions | 12 months
The proportion of infusions with temporally associated adverse events (AEs) that occur during or within 1 hour, 24 hours, and 72 hours following an infusion of investigational product | 12 months
  AEs that occur during or within 1 hour, 24 hours, and 72 hours following each infusion during 12 months of the study period

SECONDARY OUTCOMES:
The Pharmacokinetic (PK) Maximum concentration of IgG subclasses | before and after 5th infusion (12 or 16 weeks)
The Pharmacokinetic (PK) Minimum concentration of IgG subclasses | before and after 5th infusion (12 or 16 weeks)
The Pharmacokinetic (PK) Half-life of IgG subclasses | before and after 5th infusion (12 or 16 weeks)
Trough serum level of IgG subclasses and specific IgG antibodies before Infusion 1 and 13 (for subjects on 28-day infusion schedule) or Infusion 1 and 17 (for subjects on 21-day infusion schedule) | 12 months
Number and proportion of subjects who failed to meet the target IgG trough level (500 mg/dL) at any time point equal to or subsequent to 5th infusion (estimated 5 half-lives) | 12 months
The overall incidence of all AEs that occur during or within 1 hour, 24 hours, and 72 hours following an infusion of investigational product | 12 months
  AEs that occur during or within 1 hour, 24 hours, and 72 hours following each infusion during 12 months of the study period
The frequency of all AEs that occur during the study regardless of the investigator's assessment of their relationship to investigational product | 13 months (12 months of treatment + 1 month of follow-up)
The frequency of suspected adverse reactions as defined by all AEs either classified as at least possibly related to GC5107 | 13 months (12 months of treatment + 1 month of follow-up)
The number and proportion of GC5107 infusions for which the infusion rate was decreased due to AEs | 12 months
The proportion of AEs considered by the investigator to be investigational product related | 13 months (12 months of treatment + 1 month of follow-up)
Viral safety (freedom from transmission of blood-borne viral diseases): the human immunodeficiency virus (HIV) type 1 & 2, hepatitis A virus (HAV), hepatitis B virus (HBV), hepatitis C virus (HCV), and parvovirus B19 | 13 months (12 months of treatment + 1 month of follow-up)

OTHER OUTCOMES:
The incidence of acute serious bacterial infections (aSBIs) defined at United States Food and Drug Administration (FDA) guidance criteria (bacterial pneumonia, bacteremia/sepsis, bacterial meningitis, visceral abscess, osteomyelitis/septic arthritis) | 13 months (12 months of treatment + 1 month of follow-up)
The incidence of infections other than acute serious bacterial infections | 13 months (12 months of treatment + 1 month of follow-up)
The number of days missed from work, school, kindergarten, day care or days unable to perform normal daily activities due to infections | 13 months (12 months of treatment + 1 month of follow-up)
The number of days that the care provider of the pediatric subject had to miss work in order to care for the child due to infections | 13 months (12 months of treatment + 1 month of follow-up)
The number of days of unscheduled physician visits due to infection | 13 months (12 months of treatment + 1 month of follow-up)
The number of days of hospitalizations due to infection | 13 months (12 months of treatment + 1 month of follow-up)
The number of days of intravenous (IV) therapeutic antibiotics | 13 months (12 months of treatment + 1 month of follow-up)
The number of days of oral (PO) therapeutic antibiotics | 13 months (12 months of treatment + 1 month of follow-up)
Time to resolution of infections | 13 months (12 months of treatment + 1 month of follow-up)
The incidence of infections by trough IgG levels | 13 months (12 months of treatment + 1 month of follow-up)
Episodes of fever (annual rate of fever episodes per subject) | 13 months (12 months of treatment + 1 month of follow-up)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (5):
  - Children's Hospital Colorado, Aurora, Colorado
  - Immunoe Health & Research Centers, Centennial, Colorado
  - Allergy Partners of North Texas Research, Dallas, Texas
  - Lysosomal and Rare Disorders Research and Treatment Center, Inc., Fairfax, Virginia
  - Children's Hospital of Richmond at VCU, Richmond, Virginia
- Bosnia and Herzegovina (2):
  - University Clinical Center Sarajevo, Sarajevo, Sarajevo
  - University clinical center Tuzla, Tuzla, Tuzla
- Institute for Child and Youth Health Care of Vojvodina, Novi Sad, Novi Sad, Serbia

IPD SHARING:
Plan to Share IPD: No